CLINICAL TRIAL: NCT06529887
Title: Evaluate the Vision / Expectations of Patients and Caregivers for Patient-Reported Experience Measures (PREMs). Single-Center Prospective Study (Calydial). Mixed Research (Quantitative and Qualitative)
Brief Title: What Does the Patient Experience Represent for Patients and Caregivers in Dialysis?
Acronym: EnquêteXP
Status: Completed | Type: Observational
Sponsor: Calydial (Other)
Collaborators: OZ'IRIS Santé (Unknown)
Responsible Party: Sponsor
Other Study IDs: Calydial enquête XP
Record Dates: First submitted 2024-07-01; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Experience, Life; Dialysis; Patient Engagement; Patient Participation; Patient Relations, Nurse; Patient Satisfaction
Keywords: patient central care; patient experience; Sharing decision making
MeSH Terms: conditions — Patient Participation; Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Dialysis patients (hemodialysis and peritoneal dialysis)
- Professionnels: Nurses and nephrologists caring for the patient

SUMMARY:
The primary objective of this work is to describe the vision, representations, and beliefs of professionals and patients regarding the role and place of the user during their care journey at the Calydial renal health facility.

Methodology: a mixed qualitative and quantitative research.

* Qualitative research: semi-structured interviews with patients and caregivers. The objective is to define the meaning of the patient experience from the perspectives of patients and caregivers.
* Single-center prospective quantitative study: design of two questionnaires (one for patients and one for caregivers). The objectives of the questionnaires are to:

  * Evaluate the feelings, experiences, and representations/beliefs of the patient experience by caregivers and patients.
  * Assess the understanding of the patient experience by caregivers and patients.
  * Compare the patient experience based on the following parameters: age of patients, gender, treatment duration, treatment location, treatment modality, patient autonomy.
  * Measure the gap between patient and caregiver perspectives to identify/adjust actions.

DETAILED DESCRIPTION:
Patient experience encompasses all interactions a healthcare organization has with a patient and their family, potentially influencing their perceptions throughout their healthcare journey. These interactions are shaped both by the policies implemented by the facility and by the personal history and culture of each patient. Patient experience is a subjective concept that can be standardized and objectified. Even if standardized, known as a care pathway, it will still be experienced differently by each patient (depending on whether they are optimistic or pessimistic, live alone or not, and whether they reside in a rural or urban area).

The objective of our work is to evaluate the experience of our care pathway, the factors influencing patient experience, and the caregiver experience. Our facility comprises several units located in the south of Lyon and the north of Isère, providing care for chronic kidney disease at all stages. Our work focused on patients with stage 5 chronic kidney disease treated with hemodialysis (center, medically assisted dialysis unit, and self-dialysis) and home dialysis (hemodialysis and peritoneal dialysis).

The primary objective of this work is to describe the vision, representations, and beliefs of professionals and patients regarding the role and place of the user during their care journey at the Calydial renal health facility.

Methodology: mixed qualitative and quantitative research.

* Qualitative research: semi-structured interviews with patients and caregivers. The objective is to define the meaning of the patient experience from the perspectives of patients and caregivers.
* Single-center prospective quantitative study: design of two questionnaires (one for patients and one for caregivers).

The objectives of the questionnaires are to:

* Evaluate the feelings, experiences, and representations/beliefs of the patient experience by caregivers and patients.
* Assess the understanding of the patient experience by caregivers and patients.
* Compare the patient experience based on the following parameters: age of patients, gender, treatment duration, treatment location, treatment modality, patient autonomy.
* Measure the gap between patient and caregiver perspectives to identify/adjust actions.

Study population The patient and caregiver questionnaires are offered to all patients and caregivers at Calydial.

Inclusions The study population will consist of hemodialysis patients agreeing to respond to the questionnaire during their visit for a dialysis session.

Inclusion criteria:

* Patient aged 18 years or older
* On hemodialysis for more than 3 months in one of the participating centers
* Regardless of the etiology of renal disease

Exclusion criteria:

* Person refusing to participate in the study
* Person unable to read or understand French well enough to complete the questionnaires
* Inability to express consent to participate in the study
* Cognitive disorders deemed incompatible with study participation by the investigator
* Psychiatric disorders deemed incompatible with study participation by the investigator
* Person protected by law
* Patient under legal protection (safeguard of justice, curatorship, and guardianship)

Study procedure This study is observational and exploratory (non-interventional research), single-center, conducted using a self-administered questionnaire via electronic tablet. The sponsor and investigators commit to conducting this research in accordance with the protocol, Good Clinical Practice guidelines, current legislative and regulatory provisions in France and internationally (particularly the General Data Protection Regulation GDPR).

The study is offered to hemodialysis patients during a dialysis session or consultation. They are informed, and their non-opposition to participation is collected. Their participation consists of:

Responding to an electronic self-assessment questionnaire on the patient experience. A caregiver can assist the patient if necessary. The questionnaire data is pseudonymized.

Providing the following information: age, gender, dialysis modality, dialysis duration, dialysis location, participation in therapeutic education.

Data collected

The quantitative questionnaire for patients will be administered on-site across all dialysis modalities. It includes 4 categories to assess:

* Patient profile (sociodemographic data)
* Patient care (dialysis experience, recognizing body reactions, considering opinions, feeling of being heard, etc.)
* Actions to be implemented (patient participation in ETP workshops, participation in working groups, access to patient associations, considering patient knowledge, etc.)
* Patient rights (user commission, user projects, patient associations, etc.) The questionnaire will be created using REDCAP software. It will then be tested with 3 patients in a medically assisted dialysis unit and 2 professionals (a clinical research associate and a dietitian). The estimated duration of the questionnaire is 20 to 30 minutes for a patient and about 15 minutes for a professional.

Data analysis An analysis of the sociodemographic and clinical characteristics of the population will be conducted. The proportion of patients included within the total eligible population will be calculated, and the characteristics (sex, age, dialysis duration) of included and eligible non-included patients will be compared to estimate the exhaustiveness and representativeness of the included population.

A descriptive analysis will be carried out to describe the sociodemographic characteristics of the respondents. Subsequently, a comparative analysis will be performed to identify the expectations, needs, and opinions of professionals and patients for quality care. Finally, a multivariate analysis will be conducted to relate sociodemographic variables to the theme of the caregiver-patient relationship.

Analyses will be performed using SAS 9.1 software. A 5% bilateral threshold will be considered for defining statistical significance.

ELIGIBILITY:
Inclusion criteria:

* Patient aged 18 years or older
* On hemodialysis for more than 3 months in one of the participating centers
* Regardless of the etiology of renal disease

Exclusion criteria:

* Person refusing to participate in the study
* Person unable to read or understand French well enough to complete the questionnaires
* Inability to express consent to participate in the study
* Cognitive disorders deemed incompatible with study participation by the investigator
* Psychiatric disorders deemed incompatible with study participation by the investigator
* Person protected by law
* Patient under legal protection (safeguard of justice, curatorship, and guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dialysis patients and professionals working at the Calydial renal health facility
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Understanding the experiences, knowledge, and patient experience | 2 years (2020 and 2021)
  Semi-structured interviews with 8 patients (all dialysis modalities) and 8 healthcare professionals to define the objectives of the quantitative survey (patient and caregiver questionnaires).
Evaluation of the care pathway experiences and factors influencing patient experience from the perspectives of patients and caregivers. | 2 months (february and march 2022)
  Quantitative questionnaires for patients (all dialysis modalities) and their caregivers (nephrologists and nurses).

CONTACTS AND LOCATIONS:
Overall Officials: Agnès CAILLETTE-BEAUDOIN, Dr, Study Director — Calydial
Locations (4):
- France (4):
  - CALYDIAL, Irigny
  - CALYDIAL, Pierre-Bénite
  - CALYDIAL, Vénissieux
  - CALYDIAL, Vienne

IPD SHARING:
Plan to Share IPD: No